CLINICAL TRIAL: NCT04549870
Title: Efficacy of Roflumilast in the Treatment of Psoriasis - a Randomised Controlled Trial
Brief Title: Efficacy of Roflumilast in the Treatment of Psoriasis
Acronym: PSORRO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Mette Gyldenløve, MD, PhD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-20013697
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Roflumilast (Active Comparator): Roflumilast 500 microgram daily (capsule)
  Interventions: Drug: Roflumilast
- Placebo (Placebo Comparator): Placebo (capsule)
  Interventions: Drug: Roflumilast

INTERVENTIONS:
Drug: Roflumilast — Treatment according to national roflumilast guidelines
  Other Names: Daxas

SUMMARY:
Roflumilast (Daxas®), a selective, long-acting inhibitor of the enzyme phosphodiesterase-4 (PDE4), is used for severe chronic obstructive pulmonary disease. Recent research suggest roflumilast is effective in treating psoriasis. The aim of this investigator-initiated trial is to study the efficacy of oral roflumilast in patients with plaque psoriasis. This has not previously been done.

DETAILED DESCRIPTION:
Aim: To investigate the efficacy of roflumilast in the treatment of psoriasis.

Design: Multicentre, double-blinded, randomised, placebo-controlled, clinical trial.

Participants: Patients ≥18 years with plaque psoriasis.

Method: Twelve weeks treatment with either roflumilast or placebo tablets. Both groups continue for an additional 12 weeks open-label treatment.

Primary endpoint: Proportion of patients achieving at least 75% reduction from baseline psoriasis area and severity index (PASI75) at week 12.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Chronic stable plaque psoriasis (min duration 6 months)
* PASI >8
* Body mass index (BMI) > 20 kg/m2
* Candidate for systemic treatment of psoriasis
* Negative pregnancy test (only women)
* Safe anticonception during entire study and at least 1 week after end of treatment (~5 times plasma half-life of roflumilast) (only applying for fertile women)

Exclusion Criteria:

* Severe immunological disease, e.g. HIV, systemic lupus, and systemic sclerosis
* Current tuberculosis
* Current viral hepatitis
* Heart failure (NYHA III-IV)
* Moderate or severe liver failure (Child-Pugh B-C)
* Current or former malignancy (basal cell carcinoma excluded)
* Current or former depression with suicidal ideation
* Topical therapy for psoriasis during within 2 of randomization or during study
* Systemic therapy for psoriasis or psoriatic arthritis within 4 weeks of randomization or during study
* Treatment with theophylline, phenobarbital, carbamazepine, or phenytoin
* Confirmed pregnancy
* Planned pregnancy within 6 months
* Breast feeding
* Blood donation during study
* Inability to complete study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
PASI75 | 12 weeks
  Proportion of patients achieving at least 75% reduction from baseline psoriasis area and severity index (PASI75) at week 12. PASI is a measure of psoriatic disease severity.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Egeberg, MD, PhD, Study Director — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baez E, Gyldenlove M, Ben Abdallah H, Emmanuel T, Sorensen JA, Thomsen SF, Zachariae C, Egeberg A, Skov L, Iversen L, Johansen C. Oral Roflumilast Suppresses Proinflammatory Cytokine Signaling and Reduces CD4+ T-Cell and Neutrophil Infiltration in Psoriasis. J Invest Dermatol. 2025 Dec;145(12):3079-3088.e3. doi: 10.1016/j.jid.2025.04.034. Epub 2025 May 20. PMID 40403838
- [Derived] Gyldenlove M, Meteran H, Sorensen JA, Fage S, Yao Y, Lindhardsen J, Nissen CV, Todberg T, Thomsen SF, Skov L, Zachariae C, Iversen L, Nielsen ML, Egeberg A. Efficacy and safety of oral roflumilast for moderate-to-severe psoriasis-a randomized controlled trial (PSORRO). Lancet Reg Health Eur. 2023 Apr 21;30:100639. doi: 10.1016/j.lanepe.2023.100639. eCollection 2023 Jul. PMID 37465323